CLINICAL TRIAL: NCT06230328
Title: Brazilian Reality of Hepatocellular Carcinoma - BRA-HEP: Multicenter Retrospective Study (Real World Evidence - RWE)
Brief Title: Brazilian Reality of Hepatocellular Carcinoma
Acronym: BRA-HEP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: D133HR00024; BRA-HEP (Other: Hospital Israelita Albert Einstein)
Record Dates: First submitted 2023-12-22; First posted 2024-01-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Carcinoma by BCLC Stage; Hepatocellular Carcinoma Stage I; Hepatocellular Carcinoma Stage II; Hepatocellular Carcinoma Stage III
Keywords: Hepatocellular carcinoma; RWE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients with early tumors at diagnosis (BCLC 0, A or B)
- Cohort 2: Pacientes com tumores avançados ao diagnóstico (BCLC C ou D)

SUMMARY:
National, multicenter, retrospective, non-randomized observational study (Real World Evidence-RWE) with the purpose of analyzing the epidemiological profile of Hepatocellular Carcinomas (BCLC A, B or C), clinical management, progression profile and overall survival of castrated patients treated in national oncology care reference centers, within the last 6 years (between 2017 to 2022).

DETAILED DESCRIPTION:
Hepatocellular carcinoma is the third leading cause of cancer-related deaths worldwide. Prognosis strongly depends of the underlying liver disease, tumor-specific characteristics such as tumor load, extrahepatic spread and portal vein branch thrombosis, as well as access to treatments. The Brazilian reality of hepatocellular tumor clinical presentation varies widely and the management profile, treatments adopted and response rates are little described. Taking into consideration the heterogeneity of health services in reference centers in Brazil, knowing the epidemiology profile and treatment of these tumors is of paramount importance to improve care for patients, deepen the knowledge in these diseases and foster for the generation of new regional researches. The primary objective of this study is to determine and describe the epidemiological profile of hepatocellular carcinoma BCLC (Barcelona Algorithm of Liver Cancer) stages 0, A, B and C of patients followed in Brazilian reference oncology centers, within the last 6 years (between 2017 to 2022). The secondary objective is to describe the treatment and endpoints patterns of 2 disease cohorts: early disease (BCLC 0, A and B) and advanced disease (BCLC C).

ELIGIBILITY:
Inclusion Criteria:

* Male and female;
* Above 18 years old;
* Hepatocellular carcinoma diagnosis (confirmed by biopsy or imaging);

Exclusion Criteria:

* Fibrollamelar carcinoma, hepatoblastoma, intrahepatic cholangiocarcinoma, neuroendocrine tumors or other less common types of liver tumors;
* Patients with incomplete staging data;
* Patients with only 1 visit to the participating site healthcare service, with loss to follow-up prior to the second visit to the participating site healthcare service;
* Previous treatment for hepatocellular carcinoma in another institution;
* Treatment with investigational drugs in a clinical trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a hepatocellular carcinoma diagnosis (early and intermediate), meeting the eligibility criteria, who have had a 1st time visit to the study sites between 2017 and 2022, and with at least 2 visits with accessible information in the medical record will be included.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Epidemiological profile and pathological staging | At first diagnosis and over 6 years (Time of retrospective observational analysis of the study)
  Identify the epidemiological profile and pathological staging of patients diagnosed with hepatocellular carcinoma treated at participating centers. Describe the treatments adopted and the response to the progression or non-progression of the disease.

SECONDARY OUTCOMES:
Description of clinical condition | At first diagnosis and over 6 years (Time of retrospective observational analysis of the study)
  Number of injuries, presence of extrahepatic disease, portal vein thrombosis and history of upper gastrointestinal bleeding, use of local therapies, type of local therapies, use of systemic therapies, progression, and conversion rate for resection or transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Diogo Bugano, Principal Investigator — Hospital Israelita Albert Einstein
Locations (11):
- Brazil (11):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Bernardo do Campo
  - Research Site, São Paulo
  - Research Site, Vitória

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HR00024&attachmentIdentifier=9de904d4-7e66-466b-a73e-2b291fdaad32&fileName=Clinical_Study_Report_(CSR)_Synopsis__PantumorHCC.pdf&versionIdentifier=